CLINICAL TRIAL: NCT05281653
Title: The Effect of Neuromuscular Training Program on Physical Fitness and Performance Components in Young Male Futsal Players
Brief Title: The Effect of Neuromuscular Training Program in Futsal Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Gülay Aras, Principal Investigator, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-10840098-772.02-788
Record Dates: First submitted 2022-03-07; First posted 2022-03-16 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Sports Physical Therapy
Keywords: futsal; neuromuscular training program; performance; physical fitness; risk of injury

STUDY DESIGN:
Intervention Model Description: Randomized controlled single-blind study
Who Masked: Outcomes Assessor
Masking Description: The person who evaluates the athletes before and after the training is blind to the study groups and training.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuromuscular Training Group (Experimental): Athletes in this group will receive progressive neuromuscular exercise training in addition to routine 2 weekly training sessions.
  Interventions: Behavioral: Neuromuscular exercise Training
- Control Group (Experimental): The routine will continue with 2 workouts per week.
  Interventions: Behavioral: Routine training sessions

INTERVENTIONS:
Behavioral: Neuromuscular exercise Training — Progressive neuromuscular exercise training
  Arms: Neuromuscular Training Group
Behavioral: Routine training sessions — Routine training sessions
  Arms: Control Group

SUMMARY:
Despite its popularity, there has been limited research on futsal, possibly due to the lack of financial interest in the game, and most of these research articles have addressed game analysis and/or physiological demands on players during match playing and training. For this reason, our aim is to evaluate the effectiveness of an 8-week neuromuscular training program on performance, physical fitness and injury risk in university futsal players.

DETAILED DESCRIPTION:
Futsal, known as five-on-five indoor soccer, is a team sport officially authorized by FIFA and is becoming more and more popular all over the world. Futsal is among the 10 risky sports with the highest traumatic injuries. Futsal-induced traumas cause undesirable consequences such as accelerated osteoarthritis, different types of injuries in the muscle-tendon region, ligament injuries, cartilage injuries, loss of physical activity and higher repetitive injuries. Activities that result in a higher level of fitness can significantly reduce the likelihood of injury and serve as a useful tool for athletes' professional careers and post-career periods.

Neuromuscular control, which is considered a critical component of motor skills, is defined as the ability to keep the body's center of gravity within the base of support. It can be categorized as static or dynamic balance and may be the most modifiable risk factor for the prevention of knee injuries. Interventions targeting neuromuscular control include dynamic lower extremity alignment during landing from a jump, shock absorption, muscle recruitment patterns; and gains improvement in balance through plyometric, strengthening, balancing, endurance and stability exercises. Neuromuscular training program can improve neuromuscular control, which can lead to improvement in balance and joint stability.

In our study, it was aimed to evaluate the effectiveness of an 8-week neuromuscular training program on performance, physical fitness and injury risk in university futsal players.

ELIGIBILITY:
Inclusion Criteria:

* Playing in Istanbul Medipol University futsal team
* 2 days a week, 2 hours training for futsal or 1 game a week and 2 hours a week, 2 days a week

Exclusion Criteria:

* History of lower extremity injury or surgery within 6 months prior to the test
* Injury three months before the study,
* Failure to heal or complete rehabilitation of previous injury,
* Physical or mental conditions that prevent them from participating in technical and tactical futsal training and/or experimental training programs
* Two or more missed training sessions

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2024-11-04 (Actual)

PRIMARY OUTCOMES:
The Tuck Jump Test | 0-8 weeks
  It is used to monitor changes in dynamic lower extremity biomechanics. In the evaluation; knee, foot, hip and jump biomechanics will be controlled over 10 parameters. Biomechanical changes during the test will be analyzed with the Kinovea program.
Horizontal Jumping Test | 0-8 weeks
  Athletes will jump as far as possible with their feet shoulder-width apart, using their arms in the horizontal direction, and the distance between the starting point and the heel of the foot will be measured and recorded
Countermovement Jumping Test | 0-8 weeks
  It will be used to test the explosive strength of the lower extremity. Participants will perform 3 vertical jumps with their hands on the hips with maximum effort and the best score will be analyzed using the Kinovea program.
Sprint Acceleration Test | 0-8 weeks
  In this test, which is used to measure the acceleration abilities of the athletes, the athletes will start from 0.3 m behind the starting line on a 10 m field and perform a linear sprint with maximum effort 2 times with a 1 minute rest. The shortest time will be kept and recorded with the stopwatch.
Repeated Sprint Test (RST) | 0-8 weeks
  The 40m RST test consists of 8x40m sprints separated by 20 seconds of passive recovery. Athletes will be asked to warm up first with a 5-minute progressive run and then to run as fast as possible between 2 lines spaced 20 m apart. The athlete will start 0.5 m behind the starting line and the times will be recorded using a stopwatch. Each participant will run 10 m from the start/finish line of the track, turn 180 degrees, then run 20 m to the other end of the track, turn 180 degrees, and finally run 10 m back from the start/finish line. After each sprint, the athletes will slow down and start ready for the next sprint. They will walk the line. Best (RSTenibest) and average sprint time (RSTort) will be recorded as performance indexes
Y Balance Test | 0-8 weeks
  In the Y balance test, the letter Y is drawn on the ground. Of the 3 determined lines, 2 back lines form an angle of 135 degrees with the front line. During the test, for the dominant and non-dominant legs, individuals try to maintain their balanced stance on one leg by reaching in 3 directions (anterior - postero-medial and postero-lateral) with each leg, and the distances reached are measured by fixing a tape measure on the floor.
Korebalance® System | 0-8 weeks
  It is a computerized balance and exercise system that offers a high-tech option for balance assessment. It has a variable air pressure system and a tilt sensor under the platform to monitor 360-degree horizontal and 20-degree vertical movements. The software of the system gives an evaluation score following the static and dynamic balance evaluations. Higher scores indicate more balance disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Gülay Aras Bayram, PhD, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)